CLINICAL TRIAL: NCT05117697
Title: Treatment of Chronic Anal Fissure by Performing a Lateral Subcutaneous Sphincterotomy.
Brief Title: Surgical Treatment of a Chronic Anal Fissure
Acronym: STCAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56IG701SSCC977
Record Dates: First submitted 2021-09-07; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Chronic Anal Fissure

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  A comparative,randomized, prospective, single-center clinical study. Patients of the main group are treated with a crack by performing a lateral subcutaneous sphincterotomy.
  In the control group, the fissure is excised in combination with a lateral subcutaneous sphincterotomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- main group (Experimental): Patients of the main group are treated with a crack by performing a lateral subcutaneous sphincterotomy.
  Interventions: Other: lateral subcutaneous sphincterotomy
- control group (Experimental): In the control group, the fissure is excised in combination with a lateral subcutaneous sphincterotomy.
  Interventions: Other: lateral subcutaneous sphincterotomy

INTERVENTIONS:
Other: lateral subcutaneous sphincterotomy — Patients of the main group are treated with a crack by performing a lateral subcutaneous sphincterotomy.
  In the control group, the fissure is excised in combination with a lateral subcutaneous sphincterotomy.

SUMMARY:
This study is aimed at studying the effectiveness and safety of surgical treatment of chronic anal fissure.

DETAILED DESCRIPTION:
A chronic anal fissure is a rupture of the mucous membrane of the anal canal, lasting more than 2 months and resistant to non-surgical treatment. This condition is accompanied by a strong pain syndrome during and after defecation (defecation). This condition is most often found in young and able-bodied adults, so the issue of treatment is of particular relevance.

The main cause of the development of a chronic anal fissure is a spasm of the internal sphincter. It should be eliminated first of all to ensure effective therapy.The investigators plan to treat a chronic anal fissure by performing a lateral subcutaneous sphincterotomy, without excision of the fissure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic anal fissure

Exclusion Criteria:

* Inflammatory diseases of the colon
* Pectenosis
* Previous surgical interventions on the anal canal
* IV grade internal and external hemorrhoids
* Rectal fistula
* Severe somatic diseases at the decompensation stage
* Pregnancy and lactation
* Anal sphincter insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Anal sphincter insufficiency | Up to 60 days
  Frequency of anal sphincter insufficiency according to the Wexner scale incontinence after the surgical intervention. Self reported daily meausure outcome, wich evaluate from 0 - to 20 points (where 0 points = full feacal continence; 20 points = full feacal incontinence).

SECONDARY OUTCOMES:
2-item pain intensity (P2) | On day 7, 30 and 60
  Self reported pain intensity after the defecation and during the day after the surgical intervention. Each item is scored 0-10 (0 = no pain; 10 = pain as bad, as can can be).
Non-Healing Wound | On day 60
  Frequency of post-operative wound epithelialization
Profilometry /sphincterometry findings | On day 30 and 60
  Internal sphincter spasm or local internal sphincter spasm by the data of anorectal profilometry / or anorectal sphincterometry
Temporary disability | Up to 60 days
  Duration of temporary disability
Relap | Up to 60 days
  Frequency of relapses

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - SSCCRussia, Moscow
  - Nikolay Goloktionov, Moscow

IPD SHARING:
Plan to Share IPD: No